CLINICAL TRIAL: NCT06283355
Title: Comparing Single Versus Repeat Parent-to-Child Nasal Microbiome Transplant on Seeding, Engraftment, and Diversity of the Neonatal Nasal Microbiome
Brief Title: Comparing Single Versus Repeat NMT on the Diversity of the Neonatal Nasal Microbiome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00433691
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Staphylococcus Aureus; Microbial Colonization; Neonatal Infection
Keywords: microbiome
MeSH Terms: conditions — Staphylococcal Infections; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single NMT (Experimental): Swab parent nares then insert swab directly into neonate nares once.
  Interventions: Biological: Nasal Microbiota Transplant (NMT)
- Repeat NMT (Experimental): Swab parents nares then insert swab directly into neonate nares multiple times.
  Interventions: Biological: Nasal Microbiota Transplant (NMT)
- Placebo (Placebo Comparator): Insert a sterile swab into neonate nares.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nasal Microbiota Transplant (NMT) — nasal microbiota transplant
  Arms: Repeat NMT; Single NMT
Biological: Placebo — Placebo sterile swab
  Arms: Placebo

SUMMARY:
This study aims to determine whether a parent-to-child nasal microbiota transplant (NMT) can seed and engraft parental organisms into the neonatal microbiome and increase the neonatal microbiome diversity.

DETAILED DESCRIPTION:
This parent-to-child NMT study will test the effect of an anterior nares, or nasal, microbiota transplant (NMT) on seeding, engraftment, and diversity of the neonatal microbiome. Neonates admitted to the Johns Hopkins Neonatal Intensive Care Unit (NICU) will be screened and parents will be approached for enrollment in the study. After consent and baseline screening of parents and neonates, eligible neonates will undergo an NMT.

ELIGIBILITY:
Inclusion Criteria:

Neonate:

1. Neonate has anticipated NICU length of stay > 7 days
2. Neonate ≥25 weeks gestation
3. At least one parent/adult provider not colonized with S. aureus (as determined by baseline screening)
4. Neonate is not colonized with S. aureus on baseline screening

Parent/Adult provider:

1. Parent/Adult provider is able to provide informed consent

Exclusion Criteria:

Neonate:

1. Neonate has had a prior clinical or surveillance culture grow S. aureus
2. Neonate is a ward of the State
3. Neonate with antenatal suspicion for immunodeficiency (e.g. sibling with known immunodeficiency, genetic syndrome with known associated immunodeficiency)
4. Neonate cannot have nasal swabs collected (due to anatomic or other clinical intervention, including nasal packing)

Parent/Adult provider:

1. Parent/adult provider had positive COVID-19 test in prior 21 days
2. Parent/adult provider with signs or symptoms of respiratory illness (e.g. runny nose, congestion, fever, cough)
3. Parent/adult provider has been in close contact with someone in the last 7 days who had a respiratory viral infection, like the cold or the flu?
4. Parent/adult provider tests positive on baseline screening test for S. aureus nasal colonization.
5. Parent/adult provider tests positive on baseline screening test for a respiratory pathogen.
6. Parent/adult provider is not able to provide written informed consent
7. Parent/adult provider is not able to be present at the bedside at the time of intervention.
8. Parent/adult provider has history of chronic sinusitis, cystic fibrosis, or an infection with a multi-drug resistant organism.
9. Inability or unwillingness to complete the Donor questionnaire or a positive response to any question on the Donor questionnaire

Ages: 0 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal nasal microbiome diversity after intervention | Day 2, 4, 7, 10, 14 days post-intervention
  This outcome will be determined by analysis of periodic surveillance swabs collected after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Milstone, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No